CLINICAL TRIAL: NCT04747834
Title: A Prospective Multicenter Study to Assess The Clinical Outcomes of Low Energy Lens Fragmentation Cataract Extraction in Patients Undergoing Cataract Surgery
Brief Title: Assessment of Low Energy Lens Fragmentation Cataract Extraction in Patients Undergoing Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MICOR-304-101
Record Dates: First submitted 2021-02-02; First posted 2021-02-10 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Subjects will be stratified into two Cohorts. Cohort 1 is comprised of eyes with mild-to- moderate cataracts only (Grade 1 to 2). Cohort 2 is comprised of eyes with moderate to more dense cataracts only (Grade 2+ to 3+).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cohort 1 (Active Comparator): Subjects with mild to moderate cataracts (Grade 1 to 2) scheduled to undergo mechanical non-phacoemulsification lens extraction using low-energy segment removal with a micro-interventional irrigation/aspiration port (MICOR-304) to evacuate the lens prior to intraocular lens insertion.
  Interventions: Device: MICOR-304
- Cohort 2 (Active Comparator): Subjects with moderate to dense cataracts (Grade 2+ to 3+) scheduled to undergo mechanical non-phacoemulsification lens extraction using low-energy segment removal with a micro-interventional irrigation/aspiration port (MICOR-304) to evacuate the lens prior to intraocular lens insertion..
  Interventions: Device: MICOR-304

INTERVENTIONS:
Device: MICOR-304 — The MICOR-304 offers a mechanical approach to lens fragmentation and aspiration which provides an alternative to phacoemulsification with no cavitation, no thermogenic energy in the eye, which can eliminate generation of heat inside the eye while maintaining the same minimally invasive surgical approach through a small clear-cornea 2.5 mm incision.

SUMMARY:
The purpose of this research study is to evaluate the clinical outcomes of the use of low-energy segment removal with a micro-interventional irrigation/aspiration port (MICOR-304) to evacuate the lens prior to intraocular lens insertion in subjects undergoing routine cataract surgery.

DETAILED DESCRIPTION:
Up to 300 eyes at up to 5 investigational sites will be enrolled in one of the two cohorts of this clinical investigation - up to 50 eyes in Cohort 1 and up to 50 eyes in Cohort 2. Only one eye per subject will be enrolled into the study. This is multicenter, multi-cohort, prospective clinical study designed to provide longitudinal, observational, non-comparative clinical outcome data for mechanical non-phacoemulsification lens extraction using low-energy segment removal with a micro-interventional irrigation/aspiration port (MICOR-304) to evacuate the lens prior to intraocular lens insertion.

Participants who meet the inclusion and exclusion will be asked to enroll in the study. The investigator or designee will explain the study purpose, procedures and responsibilities to the potential participant and provide sufficient opportunity to ask questions, while allowing adequate time for consideration of the information provided. Upon participant confirmation of interest, written informed consent will be obtained and the subject will be enrolled in the study. One copy of the informed consent document (ICD) will be retained with the subject's medical records and one copy will be provided to the subject.

Study subjects will be stratified into two Cohorts. Cohort 1 is comprised of eyes with mild-to- moderate cataracts only (Grade 1 to 2). Cohort 2 is comprised of eyes with moderate to more dense cataracts only (Grade 2+ to 3+).

Subjects will be seen at the screening visit, intraoperative visit, and at post-operative days 1, 7, and 30.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand study requirements, willing to follow study instructions and willing to return for required study follow-up visits
2. Willing and able to understand and complete the informed consent document
3. Subjects with a cataract grade of 1 to 3+ and are scheduled to undergo cataract surgery
4. Subjects ≥ 18 years of age
5. Clear intraocular media, other than cataract

Exclusion Criteria:

1. Polar cataracts
2. Zonular instability
3. History of dry eye treatments/devices and or dry eye medications other than artificial tears.
4. Concurrent participation or participation in any clinical trial up to 30 days prior to preoperative visit
5. Subjects that are pregnant, lactating or planning to become pregnant during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farrell C. Tyson, M.D., Principal Investigator — Argus Research at Cape Coral Eye Center; Young H. Choi, M.D., Principal Investigator — Young H Choi Eye Surgery Center
Locations (3):
- United States (3):
  - Young H. Choi Eye Surgery Center, Vestavia Hills, Alabama
  - Argus Research at Cape Coral Eye Center, Cape Coral, Florida
  - Chu Vision Institute, Bloomington, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in January of 2021 and was completed in January 2022. The study had remained opened since January 2022 and was going to continue recruitment eventually. It was decided by the study sponsor to not enroll any more subjects and close out the study in February of 2024. Three clinical sites participated in the study.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 44 | 56
Completed | 44 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 44 | 56 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 9 | 29
  >=65 years | 24 | 47 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (6.6) | 70.2 (6.2) | 68.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 30 | 56
  Male | 18 | 26 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 43 | 54 | 97
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 36 | 53 | 89
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 44 | 56 | 100

OUTCOME MEASURES:

1. Primary Outcome: Total Lens Removal Time
Description: Total lens removal time is defined in two phases:
  * The beginning time starts when the surgeon enters the eye with the MICOR-304 to start the lens removal process and completing when the surgeon finishes the nucleus lens removal with the MICOR-304 before changing over to irrigation and aspiration.
  * The second phase of lens removal time is the irrigation and aspiration stage for cortex removal which starts when the irrigation and aspiration tip enters the eye and completion time is when the cortex is removed.
  The total lens removal time as defined above is recorded in minutes and seconds.
Time Frame: Assessed during the surgical procedure, measured in seconds.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
seconds | 76.0 [62.0 to 90.0] | 80.1 [66.1 to 94.1]

2. Primary Outcome: Amount of Irrigation Solution Fluid Volume Used During the Surgical Procedure
Description: Total irrigation solution volume will be recorded using the indicators on the bag which will have labels that have pre-defined markers to indicate milliliters (ml) of volume of irrigation solution used for the surgical procedure.
Time Frame: Assessed during the surgical procedure, approximately 8 - 10 minutes.
Measure: Mean (95% Confidence Interval); unit: Milliliters
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Milliliters | 40.7 [36.0 to 45.3] | 35.3 [30.6 to 40.0]

3. Secondary Outcome: Total Surgical Procedure Time
Description: Total Surgical Procedure Time time is defined as the beginning time when the surgeon makes the first incision in the eye and completion time is when the eye speculum is removed at the end of the procedure. Total surgical procedure time is recorded in minutes and seconds.
Time Frame: Assessed during the surgical procedure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
seconds | 486.3 (151.7) | 440.0 (143.1)

4. Secondary Outcome: UCVA at 1-Day
Description: Assessment of subjects uncorrected visual acuity (UCVA) at day 1 postoperative. Visual acuity is assessed by the healthcare provider without the aid of glasses or spectacles.
Time Frame: Postoperative 1 Day
Population: Some outcome measures are based on participants while other outcome measures are based on means on a unit scale
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  UCVA 20/20 @ 1-Day | 14 | 15
  UCVA 20/25 @ 1-Day | 13 | 10
  UCVA 20/30 @ 1-Day | 7 | 8
  UCVA 20/40 @ 1-Day | 4 | 8
  UCVA 20/50 @ 1-Day | 3 | 2
  UCVA 20/60 @ 1-Day | 0 | 2
  UCVA 20/70 @ 1-Day | 0 | 5
  UCVA 20/80 @ 1-Day | 1 | 0
  UCVA 20/100 @ 1-Day | 0 | 1
  UCVA 20/150 @ 1-Day | 2 | 0
  UCVA 20/200 @ 1-Day | 0 | 3
  UCVA 20/320 @ 1-Day | 0 | 1
  Finger Count @ 1-Day | 0 | 1

5. Secondary Outcome: BCDVA at 1 Week
Description: Assessment of best-corrected distance visual acuity (BCDVA) at the 1-week postoperative visit. BCDVA is assessed by the healthcare provider and is a measurement of how well someone can see at 6m with corrective lenses, such as glasses or contact lenses.
Time Frame: 1- week postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 43 | 55
Participants
  Postoperative 1-Week BCDVA 20/15 | 1 | 0
  Postoperative 1-Week BCDVA 20/20 | 30 | 36
  Postoperative 1-Week BCDVA 20/25 | 10 | 11
  Postoperative 1-Week BCDVA 20/30 | 2 | 6
  Postoperative 1-Week BCDVA 20/50 | 0 | 1
  Postoperative 1-Week BCDVA 20/150 | 0 | 1

6. Secondary Outcome: BCDVA at 1 Month
Description: Assessment of BCDVA at the 1 Month postoperative visit
Time Frame: 1 month postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 43 | 55
Participants
  Postoperative 1-Month BCDVA 20/15 | 2 | 3
  Postoperative 1-Month BCDVA 20/20 | 31 | 35
  Postoperative 1-Month BCDVA 20/25 | 8 | 10
  Postoperative 1-Month BCDVA 20/30 | 1 | 6
  Postoperative 1-Month BCDVA 20/40 | 1 | 1

7. Secondary Outcome: Change in Corneal Thickness
Description: Assessment in the mean change in corneal thickness from baseline exam through the end of the study. Corneal thickness is measured using pachymetry presented with unit of measure "μm".
Time Frame: Measured at Baseline, 1 Day, 1 Week and 1 Month postoperative.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
μm
  Preoperative Corneal Thickness | 542.9 (30.8) | 540.2 (29.7)
  1 Day Corneal Thickness | 620.5 (108.2) | 641.1 (210.4)
  1 Week Corneal Thickness | 559.4 (43.6) | 563.0 (43.5)
  1 Month Corneal Thickness | 549.1 (40.2) | 543.1 (32.1)

8. Secondary Outcome: Corneal Edema
Description: Corneal edema will be assessed as the following: 0=None, 1+=Mild, 2+=Moderate and 3+=Severe
Time Frame: Pre-operative
Population: Preoperative Corneal Edema
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  0 Corneal Edema | 44 | 56
  Corneal Edema >0 | 0 | 0

9. Secondary Outcome: Corneal Edema 1 Day Postoperative
Description: Corneal edema will be assessed as the following: 0=None, 1+=Mild, 2+=Moderate, 3+=Severe
Time Frame: 1 Day Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Postoperative 1-Day No Corneal Edema | 27 | 18
  Postoperative 1-Day Mild Corneal Edema | 8 | 19
  Postoperative 1-Day Moderate Corneal Edema | 8 | 16
  Postoperative 1-Day Severe Corneal Edema | 1 | 3

10. Secondary Outcome: Corneal Edema 1-Week Postoperative
Description: Corneal edema will be assessed as the following: 0=None, 1+=Mild, 2+=Moderate, 3+=Severe
Time Frame: 1-Week Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Postoperative 1-Week No Corneal Edema | 43 | 53
  Postoperative 1-Week Mild Corneal Edema | 1 | 2
  Postoperative 1-Week Severe Corneal Edema | 0 | 1

11. Secondary Outcome: Corneal Edema 1 Month Postoperative
Description: Corneal edema will be assessed as the following: 0=None, 1+=Mild, 2+=Moderate and 3+=Severe
Time Frame: 1 Month Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 43 | 55
Participants
  No Corneal Edema | 43 | 55
  > 0 Corneal Edema | 0 | 0

12. Secondary Outcome: Corneal Cells
Description: Corneal cells will be assessed as the following: 0=>1 cell, 0.5+=1-5 cells, 1+=6-15 cells, 2+=16-25 cells, 3+=26-50 cells and 4+=>50 cells.
Time Frame: Pre-operative
Population: Preoperative >1 Corneal Cells
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  0 Corneal Cells | 44 | 56
  > 0 Corneal Cells | 0 | 0

13. Secondary Outcome: Corneal Cells
Description: as for outcome 12
Time Frame: 1 Day Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Postoperative 1 Day >1 Corneal Cells | 10 | 15
  Postoperative 1 Day 1-5 Corneal Cells | 15 | 9
  Postoperative 1 Day 6-15 Corneal Cells | 17 | 28
  Postoperative 1 Day 16-25 Corneal Cells | 1 | 4
  Postoperative 1 Day 26-50 Corneal Cells | 1 | 0

14. Secondary Outcome: Corneal Cells
Description: as for outcome 12
Time Frame: 1-Week Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Postoperative 1-Week >1 Corneal Cell | 38 | 47
  Postoperative 1-Week 1-5 Corneal Cells | 3 | 7
  Postoperative 1-Week 6-15 Corneal Cells | 3 | 2

15. Secondary Outcome: Corneal Cells
Description: as for outcome 12
Time Frame: 1-Month Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 43 | 55
Participants
  Postoperative 1-Month 0 Corneal Cells | 43 | 55
  Postoperative 1-Month >1 Corneal Cells | 0 | 0

16. Secondary Outcome: Anterior Chamber Flare
Description: Anterior chamber flare will be assessed as the following: 0-None, 1+=Faint, 2+=Moderate, (iris and lens details clear), 3+=Marked (iris and lens details hazy), 4+=Intense fibrin or plastic aqueous.
Time Frame: Pre-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Preoperative 0 Anterior Chamber Flare | 44 | 56
  Preoperative >0 Anterior Chamber Flare | 0 | 0

17. Secondary Outcome: Anterior Chamber Flare
Description: as for outcome 16
Time Frame: 1-Day Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Postoperative 1 Day 0 Anterior Chamber Flare | 41 | 51
  Postoperative 1 Day Faint Anterior Chamber Flare | 3 | 5

18. Secondary Outcome: Anterior Chamber Flare
Description: as for outcome 16
Time Frame: 1-Week Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Postoperative 1 Week 0 Anterior Chamber Flare | 44 | 56
  Postoperative 1 Week >0 Anterior Chamber Flare | 0 | 0

19. Secondary Outcome: Anterior Chamber Flare
Description: as for outcome 16
Time Frame: 1-Month Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 43 | 55
Participants
  Postoperative 1 Month 0 Anterior Chamber Flare | 43 | 55
  Postoperative 1 Month >0 Anterior Chamber Flare | 0 | 0

20. Secondary Outcome: Posterior Capsule Opacification
Description: Posterior capsule opacification will be assessed as the following: none, minimal, mild, moderate and severe.
Time Frame: Pre-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Preoperative 0 Posterior Capsule Opacification | 44 | 56
  Preoperative >0 Posterior Capsule Opacification | 0 | 0

21. Secondary Outcome: Posterior Capsule Opacification
Description: Posterior capsule opacification will be assessed as the following: none, minimal, mild, moderate and severe.
Time Frame: 1-Day Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Postoperative 1 Day 0 Posterior Capsule Opacification | 44 | 56
  Postoperative 1 Day >0 Posterior Capsule Opacification | 0 | 0

22. Secondary Outcome: Posterior Capsule Opacificaiton
Description: Posterior capsule opacification will be assessed as the following: none, minimal, mild, moderate and severe.
Time Frame: 1-Week Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Postoperative 1 Week 0 Posterior Capsule Opacification | 43 | 56
  Postoperative 1 Week Minimal Posterior Capsule Opacification | 1 | 0

23. Secondary Outcome: Posterior Capsule Opacification
Description: Posterior capsule opacification will be assessed as the following: none, minimal, mild, moderate and severe.
Time Frame: 1-Month Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 43 | 55
Participants
  Postoperative 1 Month 0 Posterior Capsule Opacification | 39 | 47
  Postoperative 1 Month Minimal Posterior Capsule Opacification | 3 | 6
  Postoperative 1 Month Mild Posterior Capsule Opacification | 1 | 1
  Postoperative 1 Month Moderate Posterior Capsule Opacification | 0 | 1

24. Secondary Outcome: Corneal Staining Erosion
Description: Corneal staining erosion will be assessed as the following: 0=None, 1+=Mild, 2+=Moderate and 3=Severe
Time Frame: Pre-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Preoperative 0 Cornea Staining Erosion | 44 | 56
  Preoperative >0 Cornea Staining Erosion | 0 | 0

25. Secondary Outcome: Corneal Staining Erosion
Description: Corneal staining erosion will be assessed as the following: 0=None, 1+=Mild, 2+=Moderate and 3=Severe
Time Frame: 1-Day Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Postoperative 1 Day 0 Cornea Staining Erosion | 43 | 54
  Postoperative 1 Day Mild Cornea Staining Erosion | 1 | 2

26. Secondary Outcome: Corneal Staining Erosion
Description: Corneal staining erosion will be assessed as the following: 0=None, 1+=Mild, 2+=Moderate and 3=Severe
Time Frame: 1-Week Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Postoperative 1 Week 0 Cornea Staining Erosion | 44 | 56
  Postoperative 1 Week >0 Cornea Staining | 0 | 0

27. Secondary Outcome: Corneal Staining Erosion
Description: Corneal staining erosion will be assessed as the following: 0=None, 1+=Mild, 2+=Moderate and 3=Severe
Time Frame: 1-Month Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 43 | 55
Participants
  Postoperative 1 Month 0 Cornea Staining | 43 | 55
  Postoperative 1 Month >0 Cornea Staining | 0 | 0

28. Secondary Outcome: Other Slit-Lamp Findings
Description: Assessment of other slit-lamp exam findings not listed on data collection form.
Time Frame: Preoperative
Population: Other slit-lamp findings mild/moderate cohort: Chalazion Right lower eyelid, Prosthesis OS, Few RK incision OU, Anterior basement membrane dystrophy, Lasik flap. Other slit-lamp findings severe cohort: Dermatochalasis, Pterygium temporal and nasal 1/2mm
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Preoperative Other Slit-Lamp Findings | 5 | 2
  Preoperative No Other Slit-Lamp Findings | 39 | 54

29. Secondary Outcome: Other Slit-Lamp Findings
Description: Assessment of other slit-lamp exam findings not listed on data collection form.
Time Frame: 1-Day Postoperative
Population: Other slit-lamp findings mild/moderate cohort: RK incisions, anterior basement membrane dystrophy, LASIK flap, Other slit-lamp findings severe cohort: Pterygium
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Postoperative 1-Day other slit-lamp findings | 3 | 1
  Postoperative 1-Day no other slit-lamp findings | 41 | 55

30. Secondary Outcome: Other Slit-Lamp Findings
Description: Assessment of other slit-lamp exam findings not listed on data collection form.
Time Frame: 1-Week Postoperative
Population: Other slit-lamp findings mild/moderate cohort: RK incisions, anterior basement membrane dystrophy, LASIK flap, Other slit-lamp findings severe cohort: Pterygium, guttata, microcystic edema.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Postoperative 1-Week Other Slit-Lamp Findings | 3 | 3
  Postoperative 1-Week No Other Slit-Lamp Findings | 41 | 53

31. Secondary Outcome: Other Slit-Lamp Findings
Description: Assessment of other slit-lamp exam findings not listed on data collection form.
Time Frame: 1-Month Postoperative
Population: Other slit-lamp findings mild/moderate cohort: Vitreous Prolapse and Suture OS, RK incisions, anterior basement membrane dystrophy, LASIK flap, corneal scar, Other slit-lamp findings severe cohort: Endothelial Crocodile Shagreen, Arcus OU, SPK, Pterygium, guttata, microcystic edema.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 43 | 55
Participants
  Postoperative 1-Month Other Slit-Lamp Findings | 6 | 5
  Postoperative 1-Month No Other Slit-Lamp Findings | 37 | 50

32. Secondary Outcome: Macula
Description: Macula is assessed as normal and abnormal with free text to specify if abnormal, assessed via dilated fundus examination.
Time Frame: Pre-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Preoperative Macula Assessment Normal | 38 | 48
  Preoperative Macula Assessment Abnormal | 6 | 8

33. Secondary Outcome: Macula
Description: as for outcome 32
Time Frame: 1-Month Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 43 | 55
Participants
  Postoperative 1-Month Macula Assessment Normal | 36 | 51
  Postoperative 1-Month Macula Assessment Abormal | 7 | 4

34. Secondary Outcome: Disc Appearance
Description: Disc appearance is assessed as normal and abnormal with free text to specify if abnormal, assessed via dilated fundus examination.
Time Frame: Pre-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Preoperative Disc Assessment Normal | 38 | 48
  Preoperative Disc Assessment Abnormal | 6 | 8

35. Secondary Outcome: Disc Appearance
Description: as for outcome 34
Time Frame: 1-Month Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 43 | 55
Participants
  Postoperative 1-Month Disc Assessment Normal | 33 | 53
  Postoperative 1-Month Disc Assessment Abnormal | 10 | 2

36. Secondary Outcome: Vessels
Description: Vessels are assessed as normal and abnormal with free text to specify if abnormal, assessed via dilated fundus examination.
Time Frame: Pre-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Preoperative Vessel Assessment Normal | 43 | 54
  Preoperative Vessel Assessment Abnormal | 1 | 2

37. Secondary Outcome: Vessels
Description: as for outcome 36
Time Frame: 1-Month Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 43 | 55
Participants
  Postoperative 1-Month Vessel Assessment Normal | 43 | 54
  Postoperative 1-Month Vessel Assessment Abnormal | 0 | 1

38. Secondary Outcome: Periphery
Description: Periphery is assessed as normal and abnormal with free text to specify if abnormal, assessed via dilated fundus examination.
Time Frame: Pre-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 44 | 56
Participants
  Preoperative Periphery Assessment Normal | 43 | 49
  Preoperative Periphery Assessment Abnormal | 1 | 7

39. Secondary Outcome: Periphery
Description: as for outcome 38
Time Frame: 1-Month Postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 43 | 55
Participants
  Postoperative 1-Month Periphery Assessment Normal | 42 | 48
  Postoperative 1-Month Periphery Assessment Abnormal | 1 | 7

ADVERSE EVENTS:
Time Frame: 1-Month
Description: Nothing more applicable
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/44 | 1/56
Other Adverse Events (participants affected / at risk) | 10/44 | 13/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=44) | Cohort 2 (N=56)
Pneumonia (Immune system disorders) | 0 (0) | 1 (1) — At 1 month postoperative (8/23/21), the subject was hospitalized with pneumonia for 3 days. The event was serious, unrelated to the study device, and the subject was released from the hospital and fully recovered.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=44) | Cohort 2 (N=56)
Study Eye - Raised IOP Requiring Treatment (Eye disorders) | 5 (5) | 7 (7) — Seven subjects had raised Intraocular Pressure (IOP) requiring treatment. All subjects recovered from the AE with no sequelae.
Study Eye - Posterior Capsule Rupture (Eye disorders) | 1 (1) | 0 (0) — During the surgical procedure, the subject had a mild posterior capsule rupture. The investigator continued with the surgery, the event resolved without sequelae and was unrelated to the study device
Study Eye -Vitreal Prolapse (Eye disorders) | 1 (1) | 0 (0) — At 1 Month Postoperative, the subject had a vitreal prolapse. At 5 months postoperative, the vitreous strand was much improved, and the subject recovered with no sequelae
Study Eye - Cystoid Macular Edema (Eye disorders) | 1 (1) | 0 (0) — At 1 month postoperative, the subject presented with cystoid macular edema. The Subject was started on Prolensa OS BID and failed to return after the study completion date.
Study Eye - Increased Inflammation (Eye disorders) | 1 (1) | 0 (0) — At 6 weeks postoperative, the subject presented with Increased Inflammation in the study eye. The subject was prescribed an NSAID and the subject recovered with no sequalae.
Study Eye - Ectropion (Eye disorders) | 1 (1) | 0 (0) — At 2 Months postoperative the subject presented with an elevated punctal mass with ectropion left lower lid. At 3 months postop the subject underwent ectropion repair with the Oculoplastics surgeon, and the ectropion had resolved.
Study Eye - Dry Eye (Eye disorders) | 1 (1) | 1 (1) — Two subjects presented with postoperative dry eye. One of the subjects had their punctal plugs replaced and the AE resolved. The other subject also had the Ectropion AE which may have caused the dry eye, the dry eye AE resolved after surgery.
Study Eye - Corneal Edema (Eye disorders) | 0 (0) | 2 (2) — Two subjects had postop corneal edema. One of the subjects was prescribed Durezol and the event resolved. The other subject no action was taken and the event resolved by the next visit.
Study Eye - Crocodile Shagreen (Eye disorders) | 0 (0) | 1 (1) — At 1 month postoperative the subject was diagnosed with a mild case of Crocodile Shagreen in both eyes which was unrelated to the study device. The subject was prescribed medication and the event resolved 2 weeks later.
Study Eye - Microcystic Corneal Edema (Eye disorders) | 0 (0) | 1 (1) — At 1 month postoperative, the subject presented with cystoid macular edema and was prescribed medication. . The subject cancelled the 2-month appointment and withdrew consent from the study. There is no further follow up for this subject.
Study Eye - IOL Exchange (Eye disorders) | 0 (0) | 1 (1) — At 5-weeks postoperative, the subject was unable to tolerate the current IOL in the study eye and had an IOL exchange. At 2 months postoperative the subject had the IOL exchange which was uneventful, and the subject recovered with no sequelae.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT04747834/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT04747834/ICF_001.pdf